CLINICAL TRIAL: NCT03077997
Title: Acceptability and Clinical Feasibility of an Internet-delivered Intervention for Psychological Distress in Patients With Type 2 Diabetes
Brief Title: Internet Intervention for Diabetes Distress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: logistics recruitment
Sponsor: Derek Richards (Other)
Collaborators: Silver Cloud Health (Other); University of Dublin, Trinity College (Other)
Responsible Party: Sponsor-Investigator, Derek Richards, Director of Clinical Research and Innovation, Silver Cloud Health
Organization: Silver Cloud Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICBTDIABETES
Record Dates: First submitted 2017-02-20; First posted 2017-03-13 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Diabetes
Keywords: Diabetes; Diabetes distress
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Space from Diabetes (Experimental): Participants will be assigned the 'Space from Diabetes' intervention in a supported mode for 8 weeks. Participants are assigned a clinical supporter, who will be a psychological well-being practitioner in an NHS Mental Health Service. As the participant works through the programme content, the supporter will provide them with a review of their progress and interactions with the platform 6 times over the 8 week supported period.
  Interventions: Behavioral: Space from Diabetes

INTERVENTIONS:
Behavioral: Space from Diabetes — Space from Diabetes is an internet-delivered cognitive behaviour therapy-based programme for symptoms of depression, anxiety, & diabetes distress in people with type 2 diabetes mellitus.

SUMMARY:
Diabetes distress is a psychological phenomenon associated with the self-management of the disease and is characterised by feelings of anxiety, guilt, helplessness, defeat, and depression. Research suggests that internet-delivered interventions have the potential to increase people's ability to self-manage their symptoms, but whether they are effective is largely unknown. This study is designed to investigate the potential effectiveness of an internet-delivered intervention for diabetes distress in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes is a chronic metabolic endocrine disorder characterised by the inability to metabolise glucose effectively. It is associated with reduced life expectancy, significant morbidity due to specific diabetes related complications, and increased risk of complications such as heart disease, stroke, and diminished quality of life. The incidence of diabetes is on the increase with approximately 347 million adults affected worldwide. Type 2 diabetes accounts for 90-95% of these cases and figures are estimated to increase to 552 million by 2030.

Lifestyle changes such as a reduction in exercise and an increase in dietary intake over the past number of years have been flagged as being responsible for this dramatic surge in the prevalence of Type 2 diabetes on a global scale.

Because diabetes is a chronic and progressive condition people not only require regular access to medical care, but the ability to self-manage symptoms on a daily basis is now considered to be an essential part of treatment. Self-management involves the continuous monitoring of dietary intake, physical activity, general health, stress levels, blood sugar levels, and adherence to medication regimens. Diabetes is a demanding illness that requires complex self-management maintenance/care on a daily basis. Coping with these demands and maintaining lifestyle changes can often be overwhelming for individuals and this can result in significant distress that includes feelings of anxiety, guilt, helplessness, defeat, and depression.

Research has demonstrated that those who display high levels of such symptoms are not necessarily clinically depressed; rather they experience high levels of emotional distress related to diabetes and their management of the disease. Diabetes distress is a distinct condition that directly relates to diabetes outcomes. It is characterised by unique emotional issues that directly relate to the burden of living with diabetes such as worry, frustration, concern and aspects of burnout.

Several factors prevent people with diabetes from accessing support and treatment for any distress they may experience in self-managing, such as poor education, personal finances, physical access to services, lack of social support, poor motivation, low self-efficacy, and negative attitudes to treatments. In addition the concept of diabetic distress is relatively new and unknown. This highlights the growing need to develop effective treatment options to overcome barriers to access for people with type 2 diabetes.

A significant amount of research in recent years has focused on diabetes self-management education and its effectiveness for improving diabetes care and glycemic control. Face-to-face lifestyle interventions with a particular focus on behaviour change are not new in the treatment and management of type 2 diabetes. In recent years, computer-based interventions have been shown to be effective for behaviour change (e.g. in smoking cessation). Researchers are now investigating whether there is a practical and cost-effective use for computer-based interventions to address more complex behaviour change such as that required in chronic disease self-management such as Type 2 diabetes .

Previous reviews of internet-delivered interventions for people with diabetes demonstrated some effects on physical and lifestyle self-management but failed to have any great impact on psychological outcomes. Previous work seems to demonstrate the need for further more integrated approaches that considers both health behaviours and their modification and behavioural health, specifically addressing significant distress that includes feelings of anxiety, guilt, helplessness, defeat, and depression. However, can an internet-delivered intervention address the self-management of diabetes through a comprehensive consideration of the distress that so often underlies the dysregulation of self-management regimes and the inevitable consequences of that? The current study seeks to begin an attempted answer by considering the clinical feasibility of a newly developed intervention called Space from Diabetes.

Design:

A mixed-method approach will be used that captures both quantitative and qualitative data. After completing screening questionnaires, eligible patients will be invited to use the intervention over an 8 week period.

Sample:

The investigators intend to recruit participants from Enfield Community Service. A sample size of 35 participants is proposed. This sample size will allow us to estimate the standard deviation of the symptom outcome measures for a future RCT.

Procedure:

Eligible patients will be invited to use the intervention over an 8 week period. The program will be advertised to patients through Enfield Community Service and GP surgeries via leaflets distributed by staff members. Participant information sheets will be administered before beginning the programme and consent forms will be obtained at the point of sign-up online. Participants can sign up online using the link provided on the leaflet to get access to the program. Participants will sign the consent form and complete screening measures online before beginning the program. Participants will then be referred to a supporter from within Enfield Community Service. Participants' post outcome measures will be gathered 8 weeks after their initial login or activation of the programme.

Ethical considerations:

Information made available to all prospective participants will inform them of exactly what is involved in participating, including the objectives of the trial and its importance. Informed consent will be obtained from each participant before they begin to use the programme. Participants will know that their involvement is voluntary and they can withdraw their participation at any time without prejudice. In order to record participant data gathered during the survey questionnaire and focus groups, participants will be fully informed about all the material that is recorded. Moreover, data will be anonymised and stored in a secure and encrypted server and retained for seven years as original source. Postal information will be collected for the purpose of participant remuneration only. This data will be kept on a separate secure and encrypted server with unique identifiers.

All materials will be submitted to appropriate ethics committee for review and approval.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25-80.
* Have type 2 diabetes for five years or more.
* Have internet access

Exclusion Criteria:

* Outside of age criteria.
* Does not have type 2 diabetes for five years or more.
* No internet access

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Diabetes Distress (As measured by the Diabetes Distress Scale) | At the end of treatment (week 8)
  Diabetes Distress Scale (DDS; Polonsky et al., 2005; Fisher et al., 2008) is a 17-item measure that focuses on 4 aspects of distress associated with diabetes: emotional burden, regimen distress, interpersonal distress and physician distress. The measure and its 4 subscales have demonstrated good internal consistency (α > .87) and convergent validity with the Center for Epidemiological Studies Depression Scale, meal planning, exercise and total cholesterol (Polonsky et al., 2005).

SECONDARY OUTCOMES:
Depression (as measured by the Patient Health Questionnaire) | At the end of treatment (week 8)
  Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001; Spitzer, Kroenke, & Williams, 1999) is a self-report measure of depression that has been widely used in screening, primary care, and research. The PHQ-9 items reflect the diagnostic criteria for depression outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) (American Psychiatric Association [APA], 2000). Summary scores range from 0-27, where larger scores reflect a greater severity of depressive symptoms. The PHQ-9 has been found to discriminated well between depressed and non-depressed individuals using the clinical cut-off of total score ≥10, with good sensitivity (88.0%), specificity (88.0%) and reliability (.89) (Kroenke et al., 2001; Spitzer et al., 1999).
Anxiety (as measured by the 7 item Generalised Anxiety Disorder inventory) | At the end of treatment (week 8)
  Generalized Anxiety Disorder-7 (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) GAD-7 comprises 7 items measuring symptoms and severity of GAD based on the DSM-IV diagnostic criteria for GAD. The GAD-7 has good internal consistency (α = .92) and good convergent validity with other anxiety scales (Spitzer et al., 2006). Higher scores indicate greater severity of symptoms. The GAD-7 has increasingly been used in large-scale studies as a generic measure of change in anxiety symptomatology, using a cut-off score of 8 (Richards & Suckling, 2009).
Work and Social Adjustment | At the end of treatment (week 8)
  Work and Social Adjustment (WASA; Mundt, Marks, Shear & Greist, 2002) is a simple, reliable and valid measure of impaired functioning. It is a simple and reliable (α >.75) 5-item self-report measure which provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships.
Satisfaction with Treatment | End of treatment (week 8)
  The Satisfaction with Treatment (SAT; Timulak & Richards, 2012) measure contains several questions that aim to assess patient satisfaction with the iCBT intervention received. The measure consists of two qualitative questions and several quantitative questions, centering on what the patients liked or disliked about the iCBT intervention.
EuroQol 5D5L | At the end of treatment (week 8)
  The EuroQol 5D5L (EQ5D5L) (Rabin, Oemar, Oppe, & on behalf of the EuroQoL Group, 2011) is a measure of health-related quality of life. The first part of the measure consists of five self-report items measuring the domains of mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each item has a possible five responses, which rank in severity (no problems - extreme problems). From these results, a societal index can be obtained, allowing for further analysis. The second part of the measure records self-reported health state on a visual analogue scale (VAS), a vertical line where the best and worst imaginable health states score 100 and 0, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — SilverCloud Health
Locations (1):
- Barnet, Enfield, and Haringey Mental Health Trust, Enfield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torpy JM, Golub RM. JAMA patient page. Diabetes. JAMA. 2011 Jun 22;305(24):2592. doi: 10.1001/jama.2011.741. No abstract available. PMID 21693751
- [Background] Feinglos, M. N., Bethel, M. A., & SpringerLink (Online service). (2008). Type 2 diabetes mellitus: An evidence-based approach to practical management. Totowa, N.J: Humana Press, a part of Springer Science+Business Media, LLC.
- [Background] Golden SH, Lazo M, Carnethon M, Bertoni AG, Schreiner PJ, Diez Roux AV, Lee HB, Lyketsos C. Examining a bidirectional association between depressive symptoms and diabetes. JAMA. 2008 Jun 18;299(23):2751-9. doi: 10.1001/jama.299.23.2751. PMID 18560002
- [Background] Powers MA, Bardsley J, Cypress M, Duker P, Funnell MM, Fischl AH, Maryniuk MD, Siminerio L, Vivian E. Diabetes self-management education and support in type 2 diabetes: a joint position statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. Diabetes Educ. 2015 Aug;41(4):417-30. doi: 10.1177/0145721715588904. Epub 2015 Jun 5. No abstract available. PMID 26047627
- [Background] Kok JL, Williams A, Zhao L. Psychosocial interventions for people with diabetes and co-morbid depression. A systematic review. Int J Nurs Stud. 2015 Oct;52(10):1625-39. doi: 10.1016/j.ijnurstu.2015.05.012. Epub 2015 Jun 6. PMID 26118440
- [Background] Grigsby AB, Anderson RJ, Freedland KE, Clouse RE, Lustman PJ. Prevalence of anxiety in adults with diabetes: a systematic review. J Psychosom Res. 2002 Dec;53(6):1053-60. doi: 10.1016/s0022-3999(02)00417-8. PMID 12479986
- [Background] Fisher L, Mullan JT, Skaff MM, Glasgow RE, Arean P, Hessler D. Predicting diabetes distress in patients with Type 2 diabetes: a longitudinal study. Diabet Med. 2009 Jun;26(6):622-7. doi: 10.1111/j.1464-5491.2009.02730.x. PMID 19538238
- [Background] Gebel, E. (2013). Diabetes distress. Diabetes Forecast. Retrieved from http://www.diabetes.org/living-with-diabetes/complications/mental-health/diabetes-distress.html
- [Background] Nam S, Chesla C, Stotts NA, Kroon L, Janson SL. Barriers to diabetes management: patient and provider factors. Diabetes Res Clin Pract. 2011 Jul;93(1):1-9. doi: 10.1016/j.diabres.2011.02.002. Epub 2011 Mar 5. PMID 21382643
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] Strine TW, Okoro CA, Chapman DP, Beckles GL, Balluz L, Mokdad AH. The impact of formal diabetes education on the preventive health practices and behaviors of persons with type 2 diabetes. Prev Med. 2005 Jul;41(1):79-84. doi: 10.1016/j.ypmed.2004.10.009. Epub 2004 Nov 19. PMID 15916996
- [Background] Franz, M. J. (2007). Lifestyle interventions across the continuum of type 2 diabetes: reducing the risks of diabetes. American Journal of Lifestyle Medicine,1(5), 327-334
- [Background] Pal K, Eastwood SV, Michie S, Farmer AJ, Barnard ML, Peacock R, Wood B, Inniss JD, Murray E. Computer-based diabetes self-management interventions for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD008776. doi: 10.1002/14651858.CD008776.pub2. PMID 23543567
- [Background] Hogan P, Dall T, Nikolov P; American Diabetes Association. Economic costs of diabetes in the US in 2002. Diabetes Care. 2003 Mar;26(3):917-32. doi: 10.2337/diacare.26.3.917. PMID 12610059
- [Background] Centers for Disease Control and Prevention. (2011). National diabetes fact sheet, 2011 Retrieved from http://www.cdc.gov/diabetes/pubs/pdf/ ndfs_2011.pdf.
- [Background] Myung SK, McDonnell DD, Kazinets G, Seo HG, Moskowitz JM. Effects of Web- and computer-based smoking cessation programs: meta-analysis of randomized controlled trials. Arch Intern Med. 2009 May 25;169(10):929-37. doi: 10.1001/archinternmed.2009.109. PMID 19468084
- [Background] Cotter AP, Durant N, Agne AA, Cherrington AL. Internet interventions to support lifestyle modification for diabetes management: a systematic review of the evidence. J Diabetes Complications. 2014 Mar-Apr;28(2):243-51. doi: 10.1016/j.jdiacomp.2013.07.003. Epub 2013 Dec 12. PMID 24332469